CLINICAL TRIAL: NCT03377972
Title: The Cohort Study of Early Esophageal Cancer or Precancerous Lesions Treated With Endoscopic Resection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2017-130
Record Dates: First submitted 2017-11-12; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Early Esophageal Cancer or Precancerous Lesions Treated With Endoscopic Resection
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WHO diagnostic standard
- Japan diagnostic standard

SUMMARY:
Endoscopic Submucosal Dissection (ESD) is currently the main method of treatment of early esophageal cancer and precancerous lesions. Therefore, the investigators are looking forward to conduct a cohort study on early esophageal cancer patients undergoing endoscopic treatment collected from Zhongshan Hospital, Fudan University, comparing the WHO standard with Japanese standard of endoscopic therapy diagnosis. In addition，the investigators will collect patients' detailed informations and analyze the risk factors for metastasis and recurrence of early esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 15-year-old
2. Undergoing endoscopic Submucosal Dissection (ESD) in ZhongShan Hospital

Exclusion Criteria:

Preoperative patients with recurrence and Lost to follow-up of patients within 1 year

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Early esophageal cancer and precancerous lesions patients undergoing endoscopic resection therapy for the first time in zhongshan hospital from September 1, 2014 to September 1,2017.
  2. Early esophageal cancer and precancerous lesions patients undergoing endoscopic resection therapy for the first time in zhongshan hospital after September 1,2017.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison WHO diagnosis standard with JAPAN in Early Esophageal Cancer patients by accessing pathological section. | December 1st,2017-December 1st,2018
  Comparison WHO diagnosis standard with JAPAN in Early Esophageal Cancer patients by accessing pathological section.